CLINICAL TRIAL: NCT05724576
Title: Intracoronary Administration of OmniMSC-AMI for Acute ST-segment Elevation Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Intervention-Phase I Clinical Trial to Assess the Safety.
Brief Title: Intracoronary Administration of OmniMSC-AMI for Acute ST-segment Elevation Myocardial Infarction Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taiwan Bio Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202002401A0
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Safety Issues
Keywords: MSC; AMI; PCI

STUDY DESIGN:
Intervention Model Description: 10 anterior wall STEMI patients without cardiogenic shock will be enrolled into group 1 (i.e., will receive 1.5 x 107 OmniMSC-AMI, n=5) and then group 2 (3.0 x 107 OmniMSC-AMI, n=5).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose allogeneic mesenchymal stromal cells (Experimental): Intracoronary administration 1.5 x 10^7 OmniMSC-AMI in first AMI patients who just underwent primary PCI
  Interventions: Biological: OmniMSC-AMI
- High dose allogeneic mesenchymal stromal cells (Experimental): Intracoronary administration 3.0 x 10^7 OmniMSC-AMI in first AMI who just underwent primary PCI
  Interventions: Biological: OmniMSC-AMI

INTERVENTIONS:
Biological: OmniMSC-AMI — 10 anterior wall STEMI patients without cardiogenic shock will be enrolled into low dose group 1 (1.5 x 10^7 OmniMSC-AMI, n=5) and then high dose group 2 (3.0 x 10^7 OmniMSC-AMI, n=5).

SUMMARY:
This study will test the hypothesis intracoronary administration of OmniMSC-AMI (allogenic bone marrow-derived mesenchymal stem cells) just after finishing the primary percutaneous coronary intervention (PCI) in ST-segment elevation myocardial infarction (STEMI) patients without cardiogenic shock is safe and may provide benefit on improving left ventricular ejection fraction (LVEF) during clinical follow-up.

DETAILED DESCRIPTION:
Despite state-of-the-art advances in the treatment of acute myocardial infarction (AMI), including early and prompt reperfusion therapy and advanced pharmaceutical therapy, AMI remains the leading cause of death of patients hospitalized for cardiovascular disease. Loss of myocardium after AMI, resulting in reducing LVEF and ultimately pump failure, are essential for unfavorable clinical outcomes and mortality, highlighting that to protect the myocardium from AMI-induced damage is the principal rule for treatment of the AMI patients. The pathological findings have clearly identified that loss of myocardium after AMI results from first ischemic necrosis, followed by ischemia-reperfusion injury, vigorous inflammatory reaction, generation of oxidative stress, and finally, upregulation of immune reaction. Thus, a phenomenon of "propagation of myocardium from injury to irrepressible death" at the moment just after AMI always occurs. These are the reasons why a satisfactory therapy for AMI is still difficult, highlighting the timing remains the Achilles' heel for salving the jeopardized myocardium. These raise the consideration of urgently to develop a new effective and safe treatment for patients.

Abundant data have shown mesenchymal stromal cells (MSC) pleiotropic capacities of anti-inflammation, immunomodulation, and tissue regeneration. Experimental studies have further demonstrated that MSC therapy effectively protected the organs from ischemic/ischemia-reperfusion injury. However, the therapeutic impact of stem cells on the clinical setting of AMI is still universally controversial. When investigators further look at the clinical trials, delayed time to apply the stem cells on AMI patients is universally consistent. Investigators have demonstrated that early intracoronary administration (i.e., at the time interval of 90 minutes after AMI induction) of OmniMSC-AMI significantly protected the left ventricular myocardium and improved LVEF in the mini-pig AMI model. The aforementioned issues and the results of our experimental study may support our hypothesis that immediate intracoronary administration of OmniMSC-AMI into the infarcted-related vessel in first AMI patients who just yet underwent primary PCI will be safe and may offer benefits in improving LVEF and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patents, with age ≤20 or ≤80 years old.
* Fit to the definition of ST-elevation myocardial infarction (anterior myocardial infarction):

  1. Chest pain onset.
  2. 12-lead EKG:V1-V6 ≥ consecutive lead ST-segment elevation ≥1 mm.
  3. TnT-I elevation.
* Into emergency ≤ 6h upon AMI presentation.
* Patients are willing to receive the treatment and sign the informed consent.

Exclusion Criteria:

* Age < 20 or >80 years old.
* History of

  1. Malignancy.
  2. Sepsis (abnormal WBC count elevation).
  3. Hematologic disorder.
  4. AIDS.
  5. Advanced liver cirrhosis.
  6. CKD stage 5 with Ccr <15 ml/min.
* AMI occurrence > 6 hours
* Non-first AMI.
* Pregnancy or breastfeeding.
* Prison.
* Cancer treatment within 2 years.
* Expected lifespan < 6 months.
* Non-suitable candidate evaluated by PI.
* Participating in other clinical trials.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days
  Number of adverse events occurring in given time frame shall be reported to evaluate overall safety.

SECONDARY OUTCOMES:
Heart function after AMI | 1-7 days
  Cardiac MRI and 2-D/3-D echo LVEF results after administration
Heart function after treatment | 6 months
  Cardiac MRI and 2-D/3-D echo LVEF results after administration

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Kan Yip, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan